CLINICAL TRIAL: NCT04247399
Title: Simulation-assisted Teaching in Learning Gastroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anders Bo Nielsen (Other)
Responsible Party: Sponsor-Investigator, Anders Bo Nielsen, Medical Doctor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OP_972
Record Dates: First submitted 2019-12-19; First posted 2020-01-30 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Endoscopy; Education; Gastroscopy; Esophagogastroduodenoscopy; Simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation-based learning + clinical training (Experimental)
  Interventions: Other: Simulation-based learning
- Clinical training (No Intervention)

INTERVENTIONS:
Other: Simulation-based learning — Pre-clinical simulation-based learning at Simbionix GI-mentor II virtual reality simulator and OGI CLA 4 phantom.
  Arms: Simulation-based learning + clinical training

SUMMARY:
This project is a single-blinded randomized controlled trial investigating the effect of simulation-based teaching in learning gastroscopy for medical doctors.

ELIGIBILITY:
Inclusion Criteria:

* Medical doctors in medical gastroenterology or surgery

Exclusion Criteria:

* prior experience with gastroscopy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Number of procedures before declared unassisted | 1 year
  Number of gastroscopies before the supervisor declare the participant ready to do unassisted upper GI endoscopies

SECONDARY OUTCOMES:
Patient satisfaction | 1 year
  Survey using "Gastrointestinal Endoscopy Satisfaction Questionnaire" a validated questionnaire using a scale from 1-5 (5 is the best).
Complication rate | 1 year
Mucosa visualization percent of the upper gastrointestinal tract | 1 year
  Assessed by endoscopy experts at video documented endoscopies
Duration of intubation | 1 year
  Duration of time that the patient is intubated with the endoscope
Time | 1 year
  Total time for the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Anders Bo Nielsen, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided